CLINICAL TRIAL: NCT06387901
Title: Dose-limiting Toxicities of Paclitaxel in Breast Cancer Patients: Studying Interactions Between Pharmacokinetics, Physical Activity, and Body Composition: an Observational Pilot Study.
Brief Title: Investigating Paclitaxel Toxicity in Breast Cancer: the Roles of Physical Activity and Body Composition.
Acronym: PABTOX
Status: Recruiting | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Vrije Universiteit Brussel (Other); University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: PABTOX - part 1
Record Dates: First submitted 2024-04-09; First posted 2024-04-29 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer; Paclitaxel Adverse Reaction; Chemotherapeutic Toxicity; Chemotherapeutic Agent Toxicity; Body Weight; Physical Inactivity
Keywords: breast cancer; chemotherapy; physical activity; body composition; muscle mass; fat mass
MeSH Terms: conditions — Breast Neoplasms; Body Weight; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples, taken within 10 minutes as well as between 16 and 26 hours post-PTX infusion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Breast Cancer Patients on Paclitaxel: Intervention: Paclitaxel Chemotherapy Generic Name: Paclitaxel Dosage Form: Intravenous infusion Dosage: 80 mg/m² Frequency: Once weekly Duration: 12 weeks
  Interventions: Drug: Paclitaxel Chemotherapy

INTERVENTIONS:
Drug: Paclitaxel Chemotherapy — Participants will receive paclitaxel, a taxane chemotherapeutic agent used in the treatment of breast cancer. The administration involves an intravenous infusion of paclitaxel at a dosage of 80 mg/m². The treatment is scheduled once a week, continuing for a total duration of 12 weeks. This regimen is part of a (neo-)adjuvant therapy for female patients diagnosed with stage II or III breast cancer. The intervention aims to assess the pharmacokinetics of paclitaxel in relation to patient body composition and physical activity, evaluating its impact on dose-limiting toxicities and overall treatment efficacy.

SUMMARY:
This study looks into how a common breast cancer treatment, paclitaxel, can sometimes cause severe side effects that make it hard for patients to continue treatment. These side effects can significantly affect a patient's quality of life and even impact their recovery and overall health costs. What's interesting about this research is that it considers how a patient's lifestyle, specifically their physical activity levels and body makeup (like how much muscle and fat they have), might influence these side effects.

The researchers are doing a detailed study with 40 women receiving paclitaxel treatment, tracking how the drug is processed in their bodies and how their body composition and physical activity might play a role in the side effects they experience. They are using a special method to monitor drug levels in the blood and are also keeping tabs on the patients' health and physical activity through questionnaires and modern tracking devices.

The goal here is twofold: first, to better understand why these side effects happen to some people and not others, and second, to develop a model that can predict who might be at higher risk for these side effects based on their body composition, lifestyle, and how their body handles the drug. This could lead to more personalized treatment plans that could help reduce the risk of severe side effects and improve the overall treatment experience for patients with breast cancer.

In simpler terms, this research is trying to find a way to make breast cancer treatment with paclitaxel safer and more comfortable by considering how a person's lifestyle and body type might affect their reaction to the drug. This could make a big difference in helping patients complete their treatment successfully and with a better quality of life.

ELIGIBILITY:
Inclusion Criteria

* Female patients with a diagnosis of breast cancer: Specifically targeting those diagnosed with stage II or III breast cancer, to understand the effects of paclitaxel within a somewhat uniform disease severity group.
* Planned for 12 cycles of Paclitaxel (PTX) in a (neo-)adjuvant setting: The study focuses on patients scheduled to undergo a standard 12-week, once-a-week paclitaxel chemotherapy regimen as part of their treatment plan.
* Age 18 or older in (pre-)menopausal status: Adult patients of any menopausal status are eligible, ensuring a wide demographic representation.
* Prior taxane use is allowed if treatment in the adjuvant setting finished over a year ago: This criterion allows for the inclusion of patients who may have previously undergone taxane-based treatments, provided there has been a sufficient washout period to minimize the influence of prior treatments on the study outcomes.

Exclusion Criteria

* Cognitive impairment (unable to understand test instructions): Ensuring participants can comprehend and follow study procedures and requirements is crucial for data integrity and participant safety.
* Participation in clinical trials of experimental drugs: To avoid confounding effects from other investigational treatments and focus on the impact of standard-of-care paclitaxel therapy.
* Documented intolerance or allergy to PTX (non-documented intolerance or allergy will lead to drop-out): Participants must be able to tolerate paclitaxel, as adverse reactions could compromise their safety and affect study results.

Interacting drugs in home medication: Patients using medications known to interact with paclitaxel could experience altered drug metabolism or increased toxicity, potentially skewing study outcomes.

* Male sex: The study is focused on breast cancer in female patients, as the disease's presentation, treatment, and outcomes can vary significantly between genders.
* Age under 18 years: Ensuring all participants are legal adults helps adhere to ethical standards and regulatory requirements concerning consent and participation in clinical research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of female patients diagnosed with stage II or III breast cancer, identified from the Medical Oncology Department of UZ Brussel, Belgium. Eligible participants are those scheduled for a standard 12-week, once-weekly paclitaxel (PTX) chemotherapy regimen in a (neo-)adjuvant setting. Inclusion criteria ensure a diverse cohort in terms of menopausal status, with prior taxane treatment permissible if concluded over a year prior. Exclusion criteria aim to maintain focus on PTX effects, excluding those with cognitive impairments, ongoing experimental drug trials, documented PTX intolerance/allergy, contraindicated medications, or males.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2025-05-06 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Identification of Body Composition Parameter (Muscle mass) Related to Dose-Limiting Toxicities (DLTs) | Assessed through the 12-week treatment period, with measurements at baseline, cycles (each cycle is 7 days), 1 (week 1), 6 (week 6), 9 (week 9), and 12 (week 12).
  This outcome measure aims to identify specific parameters related to the body composition (muscle mass (Kg)) that influence the occurrence and severity of dose-limiting toxicities in breast cancer patients undergoing paclitaxel treatment.
Identification of Body Composition Parameters (Fat %) Related to Dose-Limiting Toxicities (DLTs) | Assessed through the 12-week treatment period, with measurements at baseline, cycles (each cycle is 7 days), 1 (week 1), 6 (week 6), 9 (week 9), and 12 (week 12).
  This outcome measure aims to identify specific parameters related to the body composition (fat (%)) that influence the occurrence and severity of dose-limiting toxicities in breast cancer patients undergoing paclitaxel treatment.
Identification of Physical Activity Parameters Related to Dose-Limiting Toxicities (DLTs) | Assessed through the 12-week treatment period, with measurements at baseline, cycles (each cycle is 7 days), 1 (week 1), 6 (week 6), 9 (week 9), and 12 (week 12).
  This outcome measure aims to identify specific parameters related to physical activity levels that influence the occurrence and severity of dose-limiting toxicities in breast cancer patients undergoing paclitaxel treatment.

SECONDARY OUTCOMES:
Paclitaxel Exposure Analysis (Cmax) | Blood samples collected and analyzed at cycles 1 (week 1), 6 (week 6), 9 (week 9), and 12 (week 12) post-paclitaxel infusion. Each cycle is 7 days.
  Evaluation of paclitaxel exposure by measuring blood serum concentrations to determine the maximum concentration remains above the threshold of 0.05 µmol/L, which is predictive of DLTs in breast cancer patients.
Paclitaxel Exposure Analysis (AUC) | Blood samples collected and analyzed at cycles 1 (week 1), 6 (week 6), 9 (week 9), and 12 (week 12) post-paclitaxel infusion. Each cycle is 7 days.
  Evaluation of paclitaxel exposure by measuring blood serum concentrations to determine the duration of time the concentration remains above the threshold of 0.05 µmol/L, which is predictive of DLTs in breast cancer patients.
Number and Type of Dose-Limiting Toxicities | DLTs recorded the week following paclitaxel infusion cycles 1, 6, 9, and 12 (each cycle is 7 days).
  Documentation and analysis of the number and type of DLTs experienced by participants, graded according to the Common Terminology Criteria for Adverse Events (CTCAE) classification v5.0. This includes monitoring for neutropenia and chemotherapy-induced peripheral neuropathy among other toxicities.

OTHER OUTCOMES:
Treatment-Related Adverse Events | During the whole treatment (12 cycles, each cycle is 7 days) and 7 days post-treatment.
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0
Body Composition Measurement via Bioelectrical Impedance Analysis (BIA) (muscle mass) | BIA assessments are scheduled at baseline (prior to the start of paclitaxel treatment), cycle 6 (week 6), and cycle 12 (week 12). Each cycle is 7 days.
  This outcome measure involves assessing muscle mass (kg), using Bioelectrical Impedance Analysis (BIA). The aim is to determine the impact of body composition on pharmacokinetics and the occurrence of dose-limiting toxicities (DLTs) in breast cancer patients undergoing paclitaxel treatment.
Body Composition Measurement via Bioelectrical Impedance Analysis (BIA) (fat %) | BIA assessments are scheduled at baseline (prior to the start of paclitaxel treatment), cycle 6 (week 6), and cycle 12 (week 12). Each cycle is 7 days.
  This outcome measure involves assessing fat %, using Bioelectrical Impedance Analysis (BIA). The aim is to determine the impact of body composition on pharmacokinetics and the occurrence of dose-limiting toxicities (DLTs) in breast cancer patients undergoing paclitaxel treatment.
Body Composition Measurement via Dual X-ray Absorptiometry (DEXA) (muscle mass) | DEXA scans are conducted at baseline (prior to the start of paclitaxel treatment), cycle 6 (week 6), and cycle 12 (week 12). Each cycle is 7 days.
  This outcome measure involves the use of Dual X-ray Absorptiometry (DEXA) to assess skeletal muscle mass (kg) in the whole body and segmented regions. This analysis aims to explore the relationship between body composition and the pharmacodynamics of paclitaxel, focusing on its efficacy and toxicity.
Body Composition Measurement via Dual X-ray Absorptiometry (DEXA) (fat mass) | DEXA scans are conducted at baseline (prior to the start of paclitaxel treatment), cycle 6 (week 6), and cycle 12 (week 12). Each cycle is 7 days.
  This outcome measure involves the use of Dual X-ray Absorptiometry (DEXA) to assess fat mass (kg) in the whole body and segmented regions. This analysis aims to explore the relationship between body composition and the pharmacodynamics of paclitaxel, focusing on its efficacy and toxicity.
Body Composition Measurement via Dual X-ray Absorptiometry (DEXA) (extracellular fluid) | DEXA scans are conducted at baseline (prior to the start of paclitaxel treatment), cycle 6 (week 6), and cycle 12 (week 12). Each cycle is 7 days.
  This outcome measure involves the use of Dual X-ray Absorptiometry (DEXA) to assess extracellular fluid (L), in the whole body and segmented regions. This analysis aims to explore the relationship between body composition and the pharmacodynamics of paclitaxel, focusing on its efficacy and toxicity.
The European Organization for Research and Treatment of Cancer quality of life questionnaire (EORTC QLQ-C30) | Administered at baseline (prior to the start of paclitaxel treatment), and after cycles 6 (week 6), 9 (week 9), and 12 (week 12). Each cycle is 7 days.
  The EORTC QLQ-C30 is a well-established instrument designed to assess the quality of life in cancer patients. It covers various dimensions including physical, emotional, and social functioning, as well as symptoms related to cancer and its treatment. This questionnaire aims to evaluate how paclitaxel treatment impacts the overall well-being and daily functioning of breast cancer patients.
EORTC QLQ-BR45 Breast (BR) Cancer Module | Completed alongside the QLQ-C30 at baseline, and following cycles 6, 9, and 12. Each cycle is 7 days.
  This questionnaire is an add-on module to the QLQ-C30 for patients with breast cancer. It assesses symptoms and side effects specific to breast cancer and its treatment, body image, sexual functioning, and future perspective. The aim is to capture the specific quality of life concerns of breast cancer patients undergoing paclitaxel treatment.
EORTC QLQ- Chemotherapy-Induced Peripheral Neuropathy (CIPN) 20 | This questionnaire is administered at baseline, and following cycles 6, 9, and 12. Each cycle is 7 days.
  The QLQ-CIPN20 is designed to assess symptoms of chemotherapy-induced peripheral neuropathy, a common side effect of paclitaxel. It evaluates sensory, motor, and autonomic symptoms related to neuropathy. This questionnaire will help quantify the extent of neuropathic side effects experienced by the patients and their impact on daily activities and quality of life.
European Health Interview Survey Physical Activity Questionnaire (EHIS PAQ) | Physical activity is monitored for 7 days following paclitaxel infusion cycles 1, 6, 9, and 12. Each cycle is 7 days.
  The EHIS PAQ is designed to gather comprehensive data on physical activity levels in various domains, including work, leisure time, and daily activities. This tool will assess changes in physical activity patterns among breast cancer patients receiving paclitaxel and explore correlations with treatment outcomes and quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Nele Adriaenssens, PhD, Principal Investigator — Vrije Universiteit Brussel
Locations (2):
- Belgium (2):
  - UZ Brussel, Brussels, Jette
  - Vrije Universiteit Brussel, Brussels, Jette

IPD SHARING:
Plan to Share IPD: Undecided
The protocol emphasizes adherence to General Data Protection Regulation (GDPR) and mentions data storage and management practices to ensure confidentiality and security. However, it does not specify arrangements for sharing IPD outside the research team or with the broader scientific community post-study.

REFERENCES:
- See also: Kom op Tegen Kanker project — https://www.komoptegenkanker.be/projecten/interacties-tussen-farmacokinetiek-van-paclitaxel-fysieke-activiteit-en-lichaamssamenstelling-bij